CLINICAL TRIAL: NCT00251095
Title: A Multicenter Phase 3, Randomized Comparison of the Safety and Efficacy of Weekly TOCOSOL(R) Paclitaxel vs. Weekly Paclitaxel Injection in the Treatment of Metastatic Breast Cancer
Brief Title: Comparison of Safety and Efficacy of TOCOSOL(R) Paclitaxel Versus Taxol(R) for Treatment of Metastatic Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Failed primary endpoint
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Monica S. Krieger, VP Regulatory Affairs, OncoGenex Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SON-8184-1075
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Breast Neoplasm
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

ARMS (2):
- Taxol (Active Comparator): Taxol 80mg/m2/week
  Interventions: Drug: Taxol
- TOCOSOL (Experimental): TOCOSOL Paclitaxel
  Interventions: Drug: TOCOSOL Paclitaxel

INTERVENTIONS:
Drug: Taxol
  Arms: Taxol
Drug: TOCOSOL Paclitaxel — 100 mg/m2/week
  Arms: TOCOSOL

SUMMARY:
The purpose of this study is to compare the objective response rates of patients randomized to receive either TOCOSOL(R) Paclitaxel or Taxol(R) (paclitaxel injection) administered every week to patients with metastatic breast cancer. The study hypothesis is that the objective response rate with TOCOSOL Paclitaxel given every week is non-inferior to that observed with Taxol given every week.

DETAILED DESCRIPTION:
Female patients with first or second line metastatic breast cancer will be randomized to receive either weekly TOCOSOL Paclitaxel or weekly Taxol (paclitaxel injection). Patients will undergo radiographic imaging of their disease to assess response to therapy. The primary endpoint of this study is a comparison of the objective response rates observed in patients receiving TOCOSOL Paclitaxel, to those receiving Taxol. Time-to-disease progression and overall survival will also be compared. The toxicities of the two treatment regimens will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic diagnosis of breast carcinoma
* Stage IV (M1) disease
* Adult (18 years of age or older) patients

Exclusion Criteria:

* Patients treated with a taxane within the past year
* Patients whose tumor tissue is known to show over expression of HER2/neu

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 821 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Objective response rates | Based on enrollment
Toxicities | Based on enrollment

SECONDARY OUTCOMES:
Median overall survival | Based on enrollment
Progression-free survival | Based on enrollment
Time-to-disease progression | Based on enrollment

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Stockton Hematology Oncology, Stockton, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mountain State Tumor Institute, Boise, Idaho
  - Oncology Care Associates, Saint Joseph, Michigan
  - Southfield Oncology Institute, Inc, Southfield, Michigan
  - Norris Cotton Cancer Center, Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Essex Oncology of North Jersey, Belleville, New Jersey
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Hematology Oncology Consultants, Inc, Columbus, Ohio
  - Chattanooga Oncology & Hematology Associates, PC, Chattanooga, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas